CLINICAL TRIAL: NCT00782197
Title: Efficacy and Safety of the Infiltration of Autologous Plasma Rich in Growth Factors (PRGF) in the Symptomatic Treatment of Knee Osteoarthritis
Brief Title: Autologous Plasma Rich in Growth Factors (PRGF) Treating the Symptomatic Knee OA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotechnology Institute IMASD (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTI-01-EC/07/ART
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Joint Disease
Keywords: osteoarthritis; knee; PRGF; autologous plasma; plasma preparations; treatment
MeSH Terms: conditions — Joint Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PRGF
  Interventions: Device: PRGF Intraarticular injection
- 2 (Active Comparator): Hyaluronic Acid
  Interventions: Device: Hyaluronic Acid Intraarticular injection

INTERVENTIONS:
Device: PRGF Intraarticular injection — Three consecutive PRGF injections each one week apart.
  Arms: 1
Device: Hyaluronic Acid Intraarticular injection — Three consecutive Hyaluronic acid (EUFLEXXA) injections, each one week apart.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PRGF infiltrations in the treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Several studies have shown the positive effects of the autologous "Preparation Rich in Growth Factors" (PRGF) in different clinical situations involving connective tissues and also in OA synovial cells. PRGF is a biological delivery system of a complex mixture of bioactive proteins essential to natural repair including anabolic factors for cartilage such as transforming growth factor-β1 (TGF-β1), platelet-derived growth factor (PDGF) and insulin-like growth factor (IGF-I). The potential of PRGF to enhance the limited capacity of cartilage to repair itself encouraged the idea of treating degenerative joint conditions with this autologous preparation.

The present study was undertaken to assess the efficacy and safety of the intra-articular injection of PRGF and to obtain useful information about the clinical effects. Since pain is the most pressing problem facing people with OA, a significant improvement in pain would indicate the potential of the proposed treatment. We will also evaluate functionality and quality of life. In addition we will examine changes in novel serum and synovial fluid biomarkers and their correlation with MRI-based parameters in a subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and aged between 40 and 72 years.
* Diagnosed with osteoarthritis of the knee by radiological image.
* Pain in the joint equal to or greater than 2.5 points in EAV.
* Radiological severity:Value in the Ahlback score 3 or less.
* Body mass index between 20 and 30.
* Possibility for observation during follow-up period.

Exclusion Criteria:

* Bilateral Gonarthrosis requiring infiltration in both knees.
* Body mass index greater than 30.
* Diagnosed polyarticular disease.
* Severe mechanical deformation.
* Previous arthroscopy in the past year.
* Intraarticular infiltration of hyaluronic acid in the last 6 months.
* Rheumatic autoimmune systemic disease.
* Poorly controlled diabetes mellitus.
* Blood alterations.
* Immunosuppressive treatments and/or coumarinics.
* Treatment with steroids for 3 months prior to its inclusion in the study.
* Treatment with nonsteroidal anti-inflammatory drugs for 15 days prior to its inclusion in the study.

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-01

PRIMARY OUTCOMES:
Improvement in Womac pain subscore and visual analogue score from baseline and changes in Lequesne's algofunctional index. | 6 months

SECONDARY OUTCOMES:
Improvement of joint function (change in Womac OA index total score and function and stiffness subscores.) | 6 months
Changes in Quality of life (SF-12 questionnaire). | 6 months
Changes in Degree of joint mobility.(determined by goniometer). | 6 months
Complications and/or adverse effects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Sanchez, Principal Investigator — UCA (Unidad de Cirugía Artroscópica Mikel Sanchez). USP Clínica la Esperanza. C/LA Esperanza 3, 01002 Vitoria (Alava)SPAIN.; Jaime Usabiaga, Study Director — Hospital Donostia; Javier Albillos, Study Director — Policlinica Gipuzkoa
Locations (3):
- Spain (3):
  - UCA (Unidad de Cirugía Artroscopica Mikel Sanchez.) Clinica USP La Esperanza., Vitoria-Gasteiz, Alava
  - Hospital Donostia., Donostia / San Sebastian, Gipuzkoa
  - Policlinica Gipuzkoa, Donostia / San Sebastian, Gipuzkoa

REFERENCES:
- See also: Related Info — http://www.prgf.net